CLINICAL TRIAL: NCT06386185
Title: Developing the Probability Algorithm for Pulmonary Hypertension Echocardiography
Acronym: DRAPE
Status: Recruiting | Type: Observational
Sponsor: Royal United Hospitals Bath NHS Foundation Trust (Other)
Collaborators: Sheffield Teaching Hospitals NHS Foundation Trust (Other); Royal Free Hospital NHS Foundation Trust (Other); Golden Jubilee National Hospital (Other Government); Papworth Hospital NHS Foundation Trust (Other Government); University of Bath (Other)
Responsible Party: Sponsor
Other Study IDs: DRAPE
Record Dates: First submitted 2024-04-23; First posted 2024-04-26 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Electrocardiography; Echocardiography; Caves

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Diagnostic Test: Patients referred for initial PH investigations, who underwent ECG and echo screening prior to RHC.
  Interventions: Diagnostic Test: Electrocardiogram; Diagnostic Test: Transthoracic echocardiogram; Diagnostic Test: Right heart catheter

INTERVENTIONS:
Diagnostic Test: Electrocardiogram — Non-invasive multi-vector voltage/time graph visualising the electrical conduction of the heart
  Other Names: ECG
Diagnostic Test: Transthoracic echocardiogram — Non-invasive 2 & 3 dimensional imaging of the heart using ultrasound
  Other Names: Echo; TTE
Diagnostic Test: Right heart catheter — Minimally invasive cardiac chamber pressure measurement using balloon catheterisation
  Other Names: RHC

SUMMARY:
The goal of this observational study is to assess the efficacy that the addition of novel markers cardiac function, particularly of right ventricular (RV) function in echocardiography, and ECG have in detecting pulmonary hypertension.

The main questions it aims to answer are:

Can novel markers in ECG and echocardiography suggest the presence of PH? Can existing screening guidelines be improved with the addition of these markers?

DETAILED DESCRIPTION:
Pulmonary Hypertension (PH) is a condition caused by high blood pressure in the blood vessels that carry blood to the lungs. It can cause severe breathlessness and failure of the right side of the heart. Sadly it is often fatal.

PH can be caused by a number of different conditions and life expectancy varies with the underlying cause, ranging from months to years. For some subtypes of PH, effective treatments exist which can significantly improve life expectancy and quality of life. Accurate tools for the assessment of PH are therefore essential, so that we can better understand and predict life expectancy and so that life-saving medications can be started earlier.

Once doctors suspect that somebody has PH, they refer them to a specialist PH centre for assessment and a procedure called right heart catheterisation (RHC), which will confirm the diagnosis. However, evidence for the suspicion of PH is frequently overlooked, leading to an average delay to diagnosis from onset of symptoms of two years. This late presentation negatively impacts survival for these patients and prevents them promptly starting the effective treatments which are available.

An electrocardiogram (ECG) is a recording of the heart's electrical signals, printed in waveforms. It is a painless, low-cost, and readily-available test used in PH assessment.

Echocardiography (echo) is a quick, safe and well-tolerated test often requested to investigate breathless patients and can provide useful information about the suspicion of PH. Echo has however been shown to lack accuracy in milder forms of the disease. It has been hypothesised that subtle markers of right ventricular function by echo, such as free wall strain (RVFWS) begin to deteriorate before the more established findings.

A large, cross-population study of ECG features and echo markers such as RVFWS both in isolation and in combination, in patients referred for PH assessment may help identify these markers, and improve detection of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18+ who have undergone TTE, ECG and RHC as part of their clinical care

Exclusion Criteria:

* Patients <18 years old
* Known or suspected congenital heart disease
* Patient has opted-out of allowing their data to be used for research and planning (via the national data opt-out choice in England, or equivalent data protection scheme in Scotland)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients aged 18+ referred for first time assessment of PH, who have undergone ECG, TTE, and RHC as part of their routine investigation.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2024-09-06 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Distinguish between patients with and without pulmonary hypertension | 2 years
  Assessment of novel echo markers of cardiac function in improving the current assessment framework's ability to correctly identify or exclude the presence of pulmonary hypertension based on a mean pulmonary artery pressure greater than 20mmHg as measured by right heart catheter.
  There is no reporting scale, rather markers will be used to assess a binary yes/no with regards to the presence of pulmonary hypertension
Distinguish between patients with pre-capillary hypertension and post-capillary hypertension | 2 years
  Assessment of novel echo markers of cardiac function in determining the subtype of pulmonary hypertension (i.e. pulmonary hypertension secondary to left heart disease, or pulmonary hypertension emanating from pulmonary abnormality) based on a mean pulmonary artery pressure greater than 20mmHg, pulmonary vascular resistance, or pulmonary capillary wedge pressure as measured by right heart catheter.
  There is no reporting scale, rather markers will be used to assess a binary yes/no with regards to the presence of pulmonary hypertension

SECONDARY OUTCOMES:
Assess the impact of the severity of pulmonary hypertension | 2 years
  Existing research has demonstrated that current assessment guidelines are less accurate in milder forms of pulmonary hypertension. We aim to assess any improvements to the overall efficacy that novel markers of cardiac function may have, particularly in those with low echocardiographic probability as determined by European Society of Cardiology echocardiographic guidelines for the assessment of pulmonary hypertension.
  There is no reporting scale, rather markers will be used to assess a binary yes/no with regards to the presence of pulmonary hypertension
Assess the impact of additional electrocardiogram markers on existing pulmonary hypertension probability stratification | 2 years
  Assessment of novel electrocardiogram markers in improving pulmonary hypertension assessment guidelines, particularly in those with low echocardiographic probability as determined by European Society of Cardiology echocardiographic guidelines for the assessment of pulmonary hypertension.
  There is no reporting scale, rather markers will be used to assess a binary yes/no with regards to the presence of pulmonary hypertension

CONTACTS AND LOCATIONS:
Overall Officials: Daniel X Augustine, Principal Investigator — Royal United Hospital
Locations (5):
- United Kingdom (5):
  - Royal United Hospital NHS Foundation Trust, Bath, Banes
  - Golden Jubilee Hospital, Glasgow, Lanarkshire
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire
  - Royal Papworth Hospital, Cambridge
  - Royal Free NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No